CLINICAL TRIAL: NCT02802670
Title: A Pharmacokinetic Study of [14C]-GDC-0810 After Single Oral Administration in Healthy Female Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: GP29916
Record Dates: First submitted 2016-05-26; First posted 2016-06-16 (Estimated); Last update posted 2016-06-16 (Estimated); Status verified 2016-06

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — 3-(4-(2-(2-chloro-4-fluorophenyl)-1-(1H-indazol-5-yl)but-1-en-1-yl)phenyl)acrylic acid

ARMS (1):
- GDC-0810 (Experimental): GDC-0810 300-mg dose administered as oral solution, containing approximately 100 microcuries of [14C]-labeled GDC-0810.
  Interventions: Drug: [14C]-GDC-0810

INTERVENTIONS:
Drug: [14C]-GDC-0810 — Participants will receive a single 300-mg dose of GDC-0810 containing approximately 100 microcuries of [14C]-labeled GDC-0810 on Day 1.
  Other Names: ARN-810; RO7056118

SUMMARY:
This is an open-label, non-randomized study to determine the excretion kinetics and mass balance of GDC-0810, and to determine metabolites present in blood, feces, and urine in healthy participants following a single 300-milligram (mg) oral dose of GDC-0810 containing approximately 100 microcuries of [14C] labeled GDC-0810 using conventional absorption, metabolism, and excretion (AME) methodology. The entire duration of the study is up to approximately 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Healthy participants with non-child bearing potential, non-pregnant, non-lactating and either post-menopausal or surgically sterile.
* Negative pregnancy test result at Screening and at Day -1.
* Body mass index of 18.5 to 29.9 kilogram per square meter.
* Healthy condition documented with no clinically significant findings from laboratory evaluations, medical history, 12-lead electrocardiograms, and vital signs.

Exclusion Criteria:

* Significant history of metabolic, allergic, dermatological, hepatic, renal, hematological, pulmonary, cardiovascular, gastric, neurological, or psychiatric disorder.
* History of significant hypersensitivity or allergy to any drug.
* Uncontrolled hypothyroidism.
* History or presence of clinically significant abnormal electrocardiogram.
* History of venous thrombosis, endometrial disorders, thrombophilic condition, inflammatory bowel disease, chronic diarrhoea, active or latent tuberculosis, and Gilbert's syndrome.
* Major surgical procedure or significant traumatic injury within 3 months prior to study participation.
* Participation in more than one other radiolabeled investigational drug study within 12 months prior to Check-in (Day -1).
* Exposure to significant radiation occuring within 12 months prior to Check-in (Day -1).
* Any acute or chronic condition that would limit the participant's ability to participate in the clinical study.
* Failure to satisfy the Investigator of fitness to participate for any other reason.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2016-05; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Cmax for [14C]-GDC-0810 | Pre-dose (0 hr), 10, 30, 45 mins, 1, 2, 3, 4, 6, 8, 12 hrs post-dose on Day 1, Day 2 (24, 36 hrs post-dose), Days 3, 4, 5, 6, and 7 post-dose
Time to maximum concentration (Tmax) for GDC-0810 | Pre-dose (0 hr), 10, 30, 45 mins, 1, 2, 3, 4, 6, 8, 12 hrs post-dose on Day 1, Day 2 (24, 36 hrs post-dose), Days 3, 4, 5, 6, and 7 post-dose
Tmax for [14C]-GDC-0810 | Pre-dose (0 hr), 10, 30, 45 mins, 1, 2, 3, 4, 6, 8, 12 hrs post-dose on Day 1, Day 2 (24, 36 hrs post-dose), Days 3, 4, 5, 6, and 7 post-dose
Area under the Concentration-Time Curve (AUC) from Hour 0 to Last Measurable Concentration (AUC0-t) for GDC-0810 | Pre-dose (0 hr), 10, 30, 45 mins, 1, 2, 3, 4, 6, 8, 12 hrs post-dose on Day 1, Day 2 (24, 36 hrs post-dose), Days 3, 4, 5, 6, and 7 post-dose
AUC0-t for [14C]-GDC-0810 | Pre-dose (0 hr), 10, 30, 45 mins, 1, 2, 3, 4, 6, 8, 12 hrs post-dose on Day 1, Day 2 (24, 36 hrs post-dose), Days 3, 4, 5, 6, and 7 post-dose
AUC Extrapolated to Infinity (AUC0-inf) for GDC-0810 | Pre-dose (0 hr), 10, 30, 45 mins, 1, 2, 3, 4, 6, 8, 12 hrs post-dose on Day 1, Day 2 (24, 36 hrs post-dose), Days 3, 4, 5, 6, and 7 post-dose
AUC0-inf for [14C]-GDC-0810 | Pre-dose (0 hr), 10, 30, 45 mins, 1, 2, 3, 4, 6, 8, 12 hrs post-dose on Day 1, Day 2 (24, 36 hrs post-dose), Days 3, 4, 5, 6, and 7 post-dose
Apparent Terminal Rate Elimination Constant for GDC-0810 | Pre-dose (0 hr), 10, 30, 45 mins, 1, 2, 3, 4, 6, 8, 12 hours post-dose on Day 1, Day 2 (24, 36 hours post-dose), Days 3, 4, 5, 6, and 7 post-dose
Maximum Observed Concentration (Cmax) for GDC-0810 | Pre-dose [0 hour (hr)], 10, 30, 45 minutes (min), 1, 2, 3, 4, 6, 8, 12 hrs post-dose on Day 1, Day 2 (24, 36 hrs post-dose), Days 3, 4, 5, 6, and 7 post-dose
Apparent Terminal Elimination Constant for [14C]-GDC-0810 | Pre-dose (0 hr), 10, 30, 45 mins, 1, 2, 3, 4, 6, 8, 12 hours post-dose on Day 1, Day 2 (24, 36 hours post-dose), Days 3, 4, 5, 6, and 7 post-dose
Apparent Terminal Elimination Half-Life (t1/2) for GDC-0810 | Pre-dose (0 hr), 10, 30, 45 mins, 1, 2, 3, 4, 6, 8, 12 hrs post-dose on Day 1, Day 2 (24, 36 hrs post-dose), Days 3, 4, 5, 6, and 7 post-dose
t1/2 for [14C]-GDC-0810 | Pre-dose (0 hr), 10, 30, 45 mins, 1, 2, 3, 4, 6, 8, 12 hrs post-dose on Day 1, Day 2 (24, 36 hrs post-dose), Days 3, 4, 5, 6, and 7 post-dose
Apparent Oral Clearance (CL/F) for GDC-0810 | Pre-dose (0 hr), 10, 30, 45 mins, 1, 2, 3, 4, 6, 8, 12 hrs post-dose on Day 1, Day 2 (24, 36 hrs post-dose), Days 3, 4, 5, 6, and 7 post-dose
Apparent Volume of Distribution (Vz/F) for GDC-0810 | Pre-dose (0 hr), 10, 30, 45 mins, 1, 2, 3, 4, 6, 8, 12 hrs post-dose on Day 1, Day 2 (24, 36 hrs post-dose), Days 3, 4, 5, 6, and 7 post-dose
Amount of Total Radioactivity Excreted in Urine Over the Sampling Interval (Aeu) for [14C]-GDC-0810 (Whenever Possible) | Pre-dose (0 hr), 0 to 12 and 12 to 24 hrs post-dose on Day 1, Days 2 (24 to 48 hrs), 3 (48 to 72 hrs), 4 (72 to 96 hrs), 5 (96 to 120 hrs), 6 (120 to 144 hrs) post-dose, and at 24-hr interval from Days 7-14 or until clinical discharge criteria met
Cumulative Aeu (Total Aeu) of [14C]-GDC-0810 (Whenever Possible) | Pre-dose (0 hr), 0 to 12 and 12 to 24 hrs post-dose on Day 1, Days 2 (24 to 48 hrs), 3 (48 to 72 hrs), 4 (72 to 96 hrs), 5 (96 to 120 hrs), 6 (120 to 144 hrs) post-dose, and at 24-hr interval from Days 7-14 or until clinical discharge criteria met
Renal Clearance (CLR) for [14C]-GDC-0810 (Whenever Possible) | Pre-dose (0 hr), 0 to 12 and 12 to 24 hrs post-dose on Day 1, Days 2 (24 to 48 hrs), 3 (48 to 72 hrs), 4 (72 to 96 hrs), 5 (96 to 120 hrs), 6 (120 to 144 hrs) post-dose, and at 24-hr interval from Days 7-14 or until clinical discharge criteria met
Percent of Total radioactivity Excreted in Urine Over Sampling (% Feu) for [14C]-GDC-0810 (Whenever Possible) | Pre-dose (0 hr), 0 to 12 and 12 to 24 hrs post-dose on Day 1, Days 2 (24 to 48 hrs), 3 (48 to 72 hrs), 4 (72 to 96 hrs), 5 (96 to 120 hrs), 6 (120 to 144 hrs) post-dose, and at 24-hr interval from Days 7-14 or until clinical discharge criteria met
Cumulative % Feu (Total % Feu) for [14C]-GDC-0810 (Whenever Possible) | Pre-dose (0 hr), 0 to 12 and 12 to 24 hrs post-dose on Day 1, Days 2 (24 to 48 hrs), 3 (48 to 72 hrs), 4 (72 to 96 hrs), 5 (96 to 120 hrs), 6 (120 to 144 hrs) post-dose, and at 24-hr interval from Days 7-14 or until clinical discharge criteria met
Amount of Total Radioactivity Excreted in Feces Over the Sampling Interval (Aef) for [14C]-GDC-0810 (Whenever Possible) | Pre-dose (0 hr), 0 to 24 hrs post-dose on Day 1, Days 2 (24 to 48 hrs), 3 (48 to 72 hrs), 4 (72 to 96 hrs), 5 (96 to 120 hrs), 6 (120 to 144 hrs) post-dose, and at 24-hr interval from Days 7-14 post-dose or until clinical discharge criteria met
Cumulative Aef (Total Aef) for [14C]-GDC-0810 (Whenever Possible) | Pre-dose (0 hr), 0 to 24 hrs post-dose on Day 1, Days 2 (24 to 48 hrs), 3 (48 to 72 hrs), 4 (72 to 96 hrs), 5 (96 to 120 hrs), 6 (120 to 144 hrs) post-dose, and at 24-hr interval from Days 7-14 post-dose or until clinical discharge criteria met
Percent of Total radioactivity Excreted in Feces Over Sampling (% Fef) for [14C]-GDC-0810 (Whenever Possible) | Pre-dose (0 hr), 0 to 24 hrs post-dose on Day 1, Days 2 (24 to 48 hrs), 3 (48 to 72 hrs), 4 (72 to 96 hrs), 5 (96 to 120 hrs), 6 (120 to 144 hrs) post-dose, and at 24-hr interval from Days 7-14 post-dose or until clinical discharge criteria met
Cumulative % Fef (Total % Fef) for [14C]-GDC-0810 (Whenever Possible) | Pre-dose (0 hr), 0 to 24 hrs post-dose on Day 1, Days 2 (24 to 48 hrs), 3 (48 to 72 hrs), 4 (72 to 96 hrs), 5 (96 to 120 hrs), 6 (120 to 144 hrs) post-dose, and at 24-hr interval from Days 7-14 post-dose or until clinical discharge criteria met

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- Madison, Wisconsin, United States